CLINICAL TRIAL: NCT05212597
Title: Multicenter, Randomized, Open-label Trial to Assess the Efficacy of Sacubitril/Valsartan vs. Amlodipine/Losartan on Left Ventricular Remodeling in Patients With Chronic Severe Aortic Regurgitation
Brief Title: Open Label RCT for Chronic Severe AR : Entresto vs. CCB/ARB
Acronym: REVERSE-AR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyoung Kim, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: reverseAR
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — sacubitril and valsartan sodium hydrate drug combination; amlodipine-losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril-Valsartan Group (Active Comparator): Participant start Sacubitril/Valsartan tablet 50mg twice a day and uptitrate to 100mg twice a day. Participants take the maximum dose considering blood pressure for a total of 48 weeks.
  Interventions: Drug: Sacubitril-valsartan
- Amlodipine-Losartan group (Placebo Comparator): Participant start amlodipine/losartan 25/2.5mg once a day and uptitrate to 5/100mg once a day. Participants take the maximum dose considering blood pressure for a total of 48 weeks.
  Interventions: Drug: Amlodipine-losartan

INTERVENTIONS:
Drug: Sacubitril-valsartan — 50mg~100mg twice daily
  Other Names: Entresto
  Arms: Sacubitril-Valsartan Group
Drug: Amlodipine-losartan — amlodipine/losartan 2.5/25mg ~ 5/100mg once daily
  Other Names: Amosartan
  Arms: Amlodipine-Losartan group

SUMMARY:
The purpose of this study is to assess the efficacy of sacubitril-valsartan compared to the combination of ARB/CCB on left ventricular remodeling in patients with chronic aortic valve regurgitation.

DETAILED DESCRIPTION:
After being informed consent about the study and potential risk, all patients giving written informed consent will undergo a 1 month screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in an open-label manner in a 1:1 ratio to sacubitril-valsartan or amlodipine/losartan.

ELIGIBILITY:
Inclusion Criteria:

1. Participant over 20 years of age who has not been hospitalized for heart failure
2. Participant with hypertension or systolic blood pressure 125 mmHg or higher
3. NYHA I
4. Participant with chronic severe aortic regurgitation (VCW >0.6cm)
5. Participant with AV regurgitant volume ≥ 60mL or effective regurgitant orifice area ≥ 0.3 cm2
6. Participant with left ventricular ejection fraction ≥ 55%

Exclusion Criteria:

1. A history of hypersensitivity or allergy to clinical trial drugs or similar compounds or ARB/NEP inhibitors
2. History of angioedema
3. Patients with an ascending aorta dilated by more than 55 mm
4. Patients with aortic valve insufficiency due to hereditary aortic disease (Marfan syndrome, Ehlers-Danlos syndrome)
5. Patients with moderate to severe aortic stenosis
6. Patients with claustrophobia or with metallic implants unsuitable for magnetic resonance imaging
7. History of acute heart failure within 6 weeks and dyspnea of NYHA II or higher
8. Symptomatic hypotension or SBP < 100 mmHg at screening
9. Patients with renal failure (Estimated GFR < 30 mL/min/1.73 m2) or on dialysis
10. Significant increase in blood potassium level (Potassium > 5 mmol/L)
11. Blood AST or ALT value is more than twice the upper limit of normal or symptoms and signs of cirrhosis (history of hepatic coma, history of esophageal varices, history of symptomatic ascites)
12. In case of acute coronary syndrome, stroke, thoracic surgery, and percutaneous coronary angioplasty within 3 months
13. If aortic valve surgery is scheduled within the next 6 months
14. In case of severe mitral valve disease
15. Patients with primary hyperaldosteronism
16. If a woman of childbearing potential has not used double contraception
17. Women who are currently pregnant or lactating
18. When it is judged that there are clinically significant abnormalities in physical examination, diagnostic examination, electrocardiogram, etc. at the time of the screening visit

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of left ventricular end-diastolic volume index from baseline to 12 months follow-up | Baseline and month 12
  Change = [LVEDV on CMR at 12 months]-[LVEDV on CMR at baseline]

SECONDARY OUTCOMES:
Change of regurgitant volume of aortic valve regurgitation from baseline to 12 months follow-up. | Baseline and month 12
  Change = [regurgitant volume at 12 months]-[regurgitant volume at baseline]
Change of EROA of aortic valve regurgitation from baseline to 12 months follow-up. | Baseline and month 12
  Measurement of regurgitant volume of AR is derived from Doppler imaging on echocardiography.
  Change = [regurgitant volume at 12 months]-[regurgitant volume at baseline]
Change of LV end-systolic volume from baseline to 12 months follow-up. | Baseline and month 12
  Change = [LVEDV at 12 months]-[LVEDV at baseline]
Holodiastolic flow reversal in the proximal abdominal aorta and descending thoracic aorta from baseline to 12 months follow-up | Baseline and month 12
  presence or absence of holodiastolic flow reversal in the proximal abdominal and descending thoracic aorta on echocardiography
Change of NT-proBNP level from baseline to 12 months follow-up. | Baseline and month 12
  Change =[NT-proBNP at 12 months]-[NTproBNP at baseline]
Aortic valve replacement or repair operation | During 12 months after enrollment
  Any surgical event for correction of AR

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kyoung Kim, MD, PhD, Principal Investigator — Heart Vascular Stroke Institute, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea